CLINICAL TRIAL: NCT04645524
Title: Phase 2 Randomized, Double Blind, Placebo-Controlled, Single-Dose, 3-Period Crossover Study to Evaluate the Efficacy of AD182, and AD504 in Obstructive Sleep Apnea
Brief Title: Crossover Trial of AD182 and AD504 in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APX-001
Record Dates: First submitted 2020-11-21; First posted 2020-11-27 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AD182 (Experimental): Oral capsule administered before bed
  Interventions: Drug: AD182; Diagnostic Test: Polysomnography
- AD504 (Experimental): Oral capsule administered before bed
  Interventions: Drug: AD504; Diagnostic Test: Polysomnography
- Placebo (Placebo Comparator): Oral capsule administered before bed
  Interventions: Drug: Placebo; Diagnostic Test: Polysomnography

INTERVENTIONS:
Drug: AD182 — Oral capsule administered before bed
  Arms: AD182
Drug: AD504 — Oral capsule administered before bed
  Arms: AD504
Drug: Placebo — Oral capsule administered before bed
  Arms: Placebo
Diagnostic Test: Polysomnography — for all arms

SUMMARY:
This is a randomized, 3-period, placebo-controlled, crossover study to examine the efficacy and safety of AD182 and AD504 versus placebo in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
The study is designed to examine the efficacy and safety of AD182 to treat obstructive sleep apnea. The study is a three-period single-dose randomized crossover design in which patients will undergo overnight polysomnographic (PSG) testing with dosing of one of the following 3 treatments: AD182, AD504, or Placebo. Participants will return 1 week after their final crossover PSG for an end of study (EOS) Visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 25 and 65 years of age, inclusive, at the time of the screening visit
* AHI 10 to 55 events/h if meets other PSG criteria

Exclusion Criteria:

* History of narcolepsy.
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control. A medication for these purposes is defined by dosage form, such that a combination antihypertensive medication is considered 1 medication
* CPAP should not be used for at least 2 weeks prior to first study PSG
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI, average number of events for every hour of sleep) | 1 night (treatment duration)
  Apnea-Hypopnea Index, AD182 and AD504 vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Corser, MD, Principal Investigator — Intrepid Research
Locations (1):
- Intrepid research, LLC, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Corser B, Eves E, Warren-McCormick J, Rucosky G. Effects of atomoxetine plus a hypnotic on obstructive sleep apnea severity in patients with a moderately collapsible pharyngeal airway. J Clin Sleep Med. 2023 Jun 1;19(6):1035-1042. doi: 10.5664/jcsm.10464. PMID 36734173